CLINICAL TRIAL: NCT04462770
Title: A 20-Week Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial of EPX-100 (Clemizole Hydrochloride) as Adjunctive Therapy in Children and Adult Participants With Dravet Syndrome (ARGUS Trial)
Brief Title: A Study of EPX-100 (Clemizole Hydrochloride) in Participants With Dravet Syndrome
Acronym: ARGUS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Epygenix (Industry)
Collaborators: Harmony Biosciences Management, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EPX-100-001; 2024-518628-57-00 (EU CTIS Number)
Record Dates: First submitted 2020-07-06; First posted 2020-07-08 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Dravet Syndrome
Keywords: Clemizole hydrochloride; Convulsive seizure; Pediatric epilepsy; Dravet syndrome
MeSH Terms: conditions — Epilepsies, Myoclonic; Seizures

STUDY DESIGN:
Intervention Model Description: Patients are randomized 1:1 to clemizole HCl (EPX-100) or placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Double-blind clemizole HCl (Experimental): Participants will receive their first dose of study drug following randomization.
  Interventions: Drug: Clemizole HCl
- Placebo (Placebo Comparator): Participants will receive their first dose of study drug following randomization.
  Interventions: Drug: Placebo
- Open-label clemizole HCl (Experimental): Eligible participants who complete the DB Period will have the option to continue in the OLE Period, during which they will receive clemizole HCL for up to 3 years.
  Interventions: Drug: Clemizole HCl; Drug: Placebo

INTERVENTIONS:
Drug: Clemizole HCl — Clemizole HCl will be administered as an oral solution.
  Other Names: EPX-100
  Arms: Double-blind clemizole HCl; Open-label clemizole HCl
Drug: Placebo — Placebo will be administered as an oral solution.
  Arms: Open-label clemizole HCl; Placebo

SUMMARY:
This is a multicenter, Phase 3, randomized, double-blind, placebo-controlled study designed to evaluate the efficacy and safety of clemizole hydrochloride (EPX-100) as adjunctive therapy in children and adult participants with Dravet syndrome (DS).

DETAILED DESCRIPTION:
This is a global, multicenter, randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy of clemizole hydrochloride as adjunctive therapy in children and adult participants with DS. The study consists of a 4-week Observational Period, a 16-week Double-Blind (DB) Period and an Open-Label Extension (OLE) Period for up to 156 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male and female participants 2 years and older at time of consent.
2. Participant or parent/legally authorized representative (LAR) willing and able to provide written informed consent, assent (if applicable) prior to initiation of any study related procedures.
3. Clinical diagnosis of DS. Participants must have seizures which are not completely controlled by AEDs with the following criteria:

   * Onset of seizures prior to 18 months of age,
   * Normal development at onset,
   * History of at least one type of countable motor seizure (CMS),
   * Brain MRI without cortical malformation (not including mild atrophy associated with the natural progression of DS),
   * Genetic mutation of the SCN1A gene must be documented.

Key Exclusion Criteria:

1. Known sensitivity, allergy, or previous exposure to clemizole HCl.
2. Exposure to any investigational drug or device <90 days prior to screening or plans to participate in another drug or device trial at any time during the study.
3. Seizures secondary to illicit drug (this includes concomitant use of tetrahydrocannabinol [THC] and nonprescription cannabidiol preparations) or alcohol use, infection, neoplasm, demyelinating disease, degenerative neurological disease, or central nervous system disease deemed progressive, metabolic illness, or progressive degenerative disease.
4. Concurrent use of lorcaserin. Note: Prior use of lorcaserin is permitted if at least 30 days have passed since the last dose.
5. Concurrent use of fenfluramine.
6. Epilepsy surgery planned during the study or epilepsy surgery within 6 months prior to Screening.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Countable Motor Seizures Per 28 Days (CMS-28) in the Titration Plus Maintenance Periods Relative to Baseline | From Baseline Period (Day 1) up to 16 weeks
  Percent change in CMS-28 from the Baseline Period through the end of the DB period.
European Union: Percent Change in Countable Motor Seizures Per 28 Days in the Maintenance Period Relative to Baseline | From maintenance period Baseline (Day 29) up to Day 85
  Percent change in CMS-28 from the Baseline Period through the end of the maintenance period.

SECONDARY OUTCOMES:
Proportion of Participants with >=50% reduction in Countable Motor Seizures Per 28 Days in the Titration Plus Maintenance Periods Relative to Baseline | From Baseline Period (Day 1) up to 16 weeks
  Proportion of participants with >=50% reduction in CMS-28 from the Baseline Period through the end of the DB Period.
European Union: Proportion of Participants with >=50% reduction in Countable Motor Seizures Per 28 Days in the Maintenance Period Relative to Baseline | From maintenance period Baseline (Day 29) up to Day 85
  Proportion of participants with >=50% reduction in CMS-28 from the Baseline Period through the end of the maintenance period.
Number of Countable Motor Seizure-free Days in the Titration Plus Maintenance Periods Relative to Baseline | From Baseline Period (Day 1) up to 16 weeks
  Number of countable motor seizure-free days from the Baseline Period through the end of the DB Period.
European Union: Number of Countable Motor Seizure-free Days in the Maintenance Period Relative to Baseline | From maintenance period Baseline (Day 29) up to Day 85
  Number of countable motor seizure-free days from the Baseline Period through the end of the maintenance period.
Clinical Global Impression of Improvement - Clinician (CGII-C) Score | Day 85
  CGII-C score at the end of the maintenance Period. This 1-item scale asks the clinician to rate how the participant's symptoms have improved or worsened relative to baseline.
Clinical Global Impression of Improvement - Participant/Caregiver (CGII-P) Score | Day 85
  CGII-C score at the end of the maintenance Period. This 1-item scale asks the clinician to rate how the participant's symptoms have improved or worsened relative to baseline.
Percent Change in All Seizures in the Titration Plus Maintenance Periods Relative to Baseline | From Baseline Period (Day 1) up to 16 weeks
  Percent change in all seizures at the end of the DB Period.
Percent Change in All Seizures in the Maintenance Period Relative to Baseline | From maintenance period Baseline (Day 29) up to Day 85
  Percent change in all seizures at the end of the maintenance period.
Incidence of Rescue Anti-epileptic Drug (AED) Use in the Titration Plus Maintenance Periods Relative to Baseline | From Baseline Period (Day 1) up to 16 weeks
  Incidence of rescue AED use as measured by the number of days on rescue AEDs from the Baseline Period through the end of the DB Period.
Incidence of Rescue Anti-epileptic Drug Use in the Maintenance Period Relative to Baseline | From maintenance period Baseline (Day 29) up to Day 85
  Incidence of rescue AED use as measured by the number of days on rescue AEDs from the Baseline Period through the end of the maintenance period.
United States FDA: Proportion of Participants with >=50% Reduction in the Countable Motor Seizures Per 28 Days in the Maintenance Period Relative to Baseline | From maintenance period Baseline (Day 29) up to Day 85
  Proportion of participants with ≥50% reduction in CMS-28 from the Baseline Period through the end of the DB Maintenance Phase only.
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From the first dose administration of study drug up to end of the study, approximately up to 172 weeks
  Incidence of TEAEs will be compared among the treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Ray, MD, Study Director — Harmony Biosciences Management, Inc.
Locations (46):
- United States (27):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California Irvine, Orange, California
  - UCSF Medical Center, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - The Nemours Foundation, Wilmington, Delaware
  - Rare Disease Research FL, Kissimmee, Florida
  - Pediatric Neurology and Epilepsy Specialists, Winter Park, Florida
  - Clinical Integrative Research Center of Atlanta (CIRCA), Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Norton Children's Research Institute, Louisville, Kentucky
  - University of Michigan- Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Nebraska, Omaha, Nebraska
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - Neurology Center for Epilepsy and Seizures, Marlboro, New Jersey
  - Weill Cornell Medical Center, New York, New York
  - Northwell Health - Lenox Hill Hospital, New York, New York
  - Duke University Health System, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Child Neurology Consultants of Austin, Austin, Texas
  - UT Southwestern/Children's Health, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Canada (4):
  - UBC Children's Hospital Research Institute, Vancouver, British Columbia
  - Children's Hospital of Eastern Ontario Research Institute Inc., Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Toronto Western Hospital, University Health Network, Toronto, Ontario
- Georgia (3):
  - Tbilisi State Medical University, Givi Zhvania Academic, Clinic of Pediatry, Tbilisi
  - Medi Club Georgia LLC, Tbilisi
  - Institute of Neurology and Neuropsychology LTD, Tbilisi
- Hungary (2):
  - Semmelweis University, Budapest
  - University of Debrecen, Debrecen
- Poland (3):
  - University Clinical Center in Gdansk, Division of Developmental Neurology, Gdansk
  - Medical Centre Plejady, Krakow
  - Institute of Mother and Child, Warsaw
- "Prof. Dr. Al. Obregia" Psychiatry Clinical Hospital, Bucharest, Romania
- Spain (2):
  - Hospital Infantil Universitario Niño Jesús, Madrid, Madrid Provincia
  - Hospital de la Santa Creu i Sant Pau, Barcelona
- United Kingdom (4):
  - Cardiff and Vale University Health Board, Cardiff
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Great Ormond Street Hospital For Children, London
  - Sheffield Children's Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No